CLINICAL TRIAL: NCT01002391
Title: Twenty-four Hours or 6 Days? A Prospective Randomized Trial Comparing Dressing Wear Time After Reduction Mammaplasty
Brief Title: Dressing Wear Time After Reduction Mammaplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Francescato Veiga (Other)
Collaborators: Universidade do Vale do Sapucai (Other)
Responsible Party: Sponsor-Investigator, Daniela Francescato Veiga, Professor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: dinter01
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Surgical Site Infection; Skin Colonization
Keywords: breast hypertrophy; mammaplasty; bandages; surgical site infection; skin colonization
MeSH Terms: conditions — Surgical Wound Infection; Gigantomastia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postoperative day 1 (Experimental): Dressing is removed on the first postoperative day
  Interventions: Procedure: reduction mammaplasty
- Postoperative day 6 (Experimental): Dressing is removed on the sixth postoperative day
  Interventions: Procedure: reduction mammaplasty

INTERVENTIONS:
Procedure: reduction mammaplasty — Dressing following reduction mammaplasty is removed on the first postoperative day
  Other Names: Breast reduction surgery
  Arms: Postoperative day 1
Procedure: reduction mammaplasty — Dressing following reduction mammaplasty is removed on the sixth postoperative day
  Other Names: Breast reduction surgery
  Arms: Postoperative day 6

SUMMARY:
This study was designed to determine whether the duration of dressing wear following reduction mammaplasty influence skin colonization and surgical site infections rates.

DETAILED DESCRIPTION:
Surgical site infections (SSI) are wound infections that occur after invasive procedures.Particularly in plastic surgery procedures, to minimize the risk of SSI is imperative, since even minor infections are able to complicate the healing process and harm the cosmetic result.

Reduction mammaplasty is an effective and well established procedure performed for the relief of physical pain and discomfort associated with macromastia, which significantly decreases patients' quality of life.Breast reduction has provided long-term relief for most patients, with high patient satisfaction.

The demand for this kind of plastic surgery is high.Reduction mammaplasty was the fifth most commonly surgical procedure performed by plastic surgeons in women of United States.Since reduction mammaplasty is associated with a high incidence of wound problems,all effort to minimize the risk of SSI is valid.

ELIGIBILITY:
Inclusion Criteria:

* breast hypertrophy
* candidate to reduction mammaplasty
* body mass index under 30Kg/m2

Exclusion Criteria:

* pregnancy, delivery or breast feeding during the last 12 months
* body mass index over 30Kg/m2
* breast cancer history
* previous breast surgery
* hard smoking

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
surgical site infection | 30 days postoperatively

SECONDARY OUTCOMES:
skin colonization | 6 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Joel Veiga-Filho, MD, MSc, Principal Investigator — Universidade do Vale do Sapucaí and Universidade Federal de São Paulo; Daniela F Veiga, MD, PhD, Study Director — Universidade do Vale do Sapucaí and Universidade Federal de São Paulo; Lydia M Ferreira, MD, PhD, Study Chair — Universidade do Vale do Sapucaí and Universidade Federal de São Paulo
Locations (1):
- Hospital das Clínicas Samuel Libânio - UNIVÁS, Pouso Alegre, Minas Gerais, Brazil

REFERENCES:
- [Result] Veiga-Filho J, Veiga DF, Sabino-Neto M, Damasceno CAV, Sales EML, Garcia ES, Oliveira IB, De Simoni LF, Juliano Y, Ferreira LM. Dressing wear time after reduction mammaplasty: a randomized controlled trial. Plast Reconstr Surg. 2012 Jan;129(1):1e-7e. doi: 10.1097/PRS.0b013e3182361ee9. PMID 22186564